CLINICAL TRIAL: NCT02393820
Title: Phase II Study of Pazopanib in Patients With Progressive Recurrent and/or Metastatic Salivary Gland Carcinoma
Brief Title: Pazopanib in Patients With Progressive Recurrent and/or Metastatic Salivary Gland Carcinoma
Acronym: PACSA-ORL02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-0130/1205; 2012-004408-36 (EudraCT Number)
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Salivary Gland Carcinoma
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pazopanib (Experimental): Pazopanib per os, 800mg daily until progression
  Interventions: Drug: pazopanib

INTERVENTIONS:
Drug: pazopanib — treatment will be given until progression or unacceptable toxicity .
  Other Names: Votrient

SUMMARY:
Open-label, multicenter, single arm phase II study, set up in collaboration with the "Réseau d'Expertise Français sur les Cancers ORL Rares" (REFCOR), evaluating the activity and safety of single agent pazopanib in recurrent or metastatic tumors in salivary gland including adenoid cystic carcinoma (ACC) and to exploring the activity and safety of pazopanib in non-adenoid cystic carcinoma (non-ACC).

DETAILED DESCRIPTION:
In the non-ACC SGCHN population, assessment of the activity of pazopanib is exploratory without a predetermined study design, with up to 20 patients. A planned interim analysis of acute toxicities was conducted 3 months after the 14th non-ACC inclusion.

ACC As the endpoint will be evaluated at 6 months after treatment start, a one-stage phase II study design was chosen. The unacceptable 6-month rate of progression free survival is 20% and the promising 6-month rate of progression free survival is 40%.

43 patients are to be treated. If ≤12 patients alive without progression at 6 months will be observed, the drug will be declared ineffective.

If ≥13 patients alive without progression at 6 months will be observed, the drug will be declared promising.

The α error rate (accepting a poor treatment) is 0.07 and the β error rate (rejecting a promising treatment) is 0.07.

Analysis of results will be separated between non ACC and ACC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of recurrent and/or metastatic salivary glands (including ACC and non ACC).
* Progressive disease within 6 months before inclusion as assessed by CT and/or MRI using at least two measurements (RECIST v1.0) with at least one measurable target lesion >10 mm.
* Recurrent and/or metastatic salivary glands carcinoma failing locoregional therapy, without possibility of curative treatment.
* Patients may have had unlimited prior therapy but must have had at least 4 weeks between any chemotherapy, radiotherapy, surgery and study enrollment.
* Tumoral tissue must be provided for subsequent histological review and biomarker analysis.
* Euthyroid patient.
* Hepatic, renal, cardiac and hematology normal functions.
* Ability to take oral medication.

Exclusion Criteria:

* Non salivary gland carcinoma (lachrymal gland tumor is excluded).
* Known or symptomatic cerebral metastasis.
* Patients treated with strong inhibitor or inductor of CYP3A4 within 14 days before inclusion.
* Presence of uncontrolled infection.
* Diagnosis of any previous malignancy within the last 5 years, except for completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma.
* Stable disease.
* Corrected QT interval (QTc) >480 msecs using Bazett's formula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-08-26 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
progression free survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joel Mr Guigay, Pr, Principal Investigator — Centre Lacassagne Nice
Locations (15):
- France (15):
  - Institut de Cancérologie de l'Ouest Paul Papin, Angers
  - CHU Bordeaux, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Centre Val d'Aurelle Paul Lamarque, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Centre Hospitalier St Joseph, Paris
  - Centre Eugène Marquis, Rennes
  - Institut Curie site St Cloud, Saint-Cloud
  - Institut Cancérologie de l'Ouest, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.